CLINICAL TRIAL: NCT06265649
Title: Acute Left Colon Diverticulitis: is it Still a Surgical Disease When Only Medical Treatment is Required? A Retrospective Study Based on Propensity Score Matching
Brief Title: Comparison of NOM for ACLD Between Medical and Surgical Ward
Status: Recruiting | Type: Observational
Sponsor: Ospedali Riuniti Trieste (Other)
Responsible Party: Principal Investigator, Manuela Mastronardi, Principal Investigator, Ospedali Riuniti Trieste
Other Study IDs: NOM-ALCD
Record Dates: First submitted 2024-01-06; First posted 2024-02-20 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Diverticulitis; Colon Disease; Acute Diverticulitis
Keywords: diverticulitis; non-operative management
MeSH Terms: conditions — Diverticulitis; Colonic Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Surgical Group (SG): Patients with ALCD undergoing NOM admitted to the surgical ward
  Interventions: Other: NOM
- Non-Surgical Group (NSG): Patients with ALCD undergoing NOM admitted to the medical ward
  Interventions: Other: NOM

INTERVENTIONS:
Other: NOM — Non-operative management (NOM) for ALCD consists of lab test monitoring, fluid therapy, antibiotic therapy, abscess drainage if >4cm, restoring a regular diet

SUMMARY:
In Europe, patients with acute left colon diverticulitis (ALCD) are usually admitted to surgical wards even when only medical treatment is required. The study compares ALCD non-operative management (NOM) between surgical and non-surgical environments regarding clinical outcomes, hospitalization length(LOS), and follow-up.

DETAILED DESCRIPTION:
Acute diverticulitis is one of the most common gastrointestinal disorders, with an estimated lifetime risk ranging from 10 to 25%. Notably this condition predominantly affects the left side of the colon (Acute Left Colon Diverticulitis - ALCD). Over the years, advancements in radiological imaging techniques have led to the modification of the original Hinchey classification, and in 2015 the World Society of Emergency Surgery (WSES) introduced a novel classification based on computer tomography (CT) findings. The prevalence of ALCD is on the rise in Western countries, with a marked increase of 132% observed between 1980 and 2007, especially among individuals aged 40 to 49 years. This trend is also evident in Italy, where there was a substantial rise in admission rates between 2008 and 2015, increasing from 8.8 to 11.8 cases per 100,000 inhabitants, primarily among those under 60 years old. Consequently, this surge in ALCD cases has led to elevated healthcare costs, particularly when surgical intervention is not required. Notably, only around 5% of patients with ALCD experience complicated episodes, indicating that uncomplicated ALCD (U-ACLD) is more common than complicated ACLD (C-ALCD). However, current clinical practice still demonstrates high admission rates for both U-ACLD and C-ALCD, particularly among the elderly with comorbidities. Given that surgery is not always warranted, patients are often admitted to non-surgical departments, although no specific guidelines exist to determine which facility is the most suitable.

There remains a dearth of knowledge regarding the comparative management of ALCD between surgical and non-surgical wards in cases of non-operative management (NOM). Some studies demonstrated similar outcomes among patients admitted to both surgical and non-surgical units.

In this context, the primary objective of the current study is to compare ALCD patients admitted for NOM to the surgical ward with those admitted to a non-surgical ward. Specifically, the study aims to assess clinical outcomes (such as gastrointestinal disorders and the restoration of a regular diet), hospitalization length (Length of Stay - LOS), and post-admission follow-up.

The following data were collected: age, sex, body mass index (BMI), American Society of Anesthesiologists (ASA) scores, previous ALCD episodes (requiring or not requiring hospitalization), C-reactive protein (CRP) levels on admission, type of management (i.e. no treatment, antimicrobial therapy, percutaneous drainage), LOS, post-discharge colonoscopy, follow-up visits, and ALCD recurrence. Follow-up data were retrieved from the electronic records covering two years after the episodes. ALCD was classified using the Hinchey classification modified by Wasvary et al. based on CT findings on admission. According to the admission department, the study population was divided into two groups: a surgical group (SG) and a non-surgical group (NSG). The ward of hospitalization was decided by the emergency doctor according to bed availability: if there were beds in the surgical ward, patients were preferably hospitalized there, otherwise, a non-surgical environment was chosen. The non-surgical wards were mainly the two wards of Internal Medicine. Criteria considered for discharge include resolution of fever, pain reduction with no need for constant use of painkillers, free oral feeding, normalization of white blood cell count, and more than a 50% decrease in the serum levels of CRP. Recurrence was defined as a new ALCD episode confirmed by a CT scan not earlier than 2 months after the first episode.

To compare ALCD management in non-surgical and surgical environments, SG subjects were propensity-score matched (PSM) to NSG subjects on ALCD grade according to the classification modified by Wasvary et al., to reduce the bias related to ALCD grade.

This decision was made also to study which factors of patients' baseline characteristics (age, sex, BMI, ASA score, CRP levels) mainly differ between the two Groups. The Shapiro-Wilk test was used to analyze quantitative variables. Nominal variables are expressed as numbers and percentages, non-normal quantitative variables as median and range, and normal variables as mean and standard deviation (SD). Chi-squared and Fisher's exact test were used to compare nominal variables, whereas the Mann-Whitney U test was used for non-normal quantitative variables and the T-student test for normal quantitative variables. A multivariate logistic regression analysis was conducted to evaluate if age, sex, ASA score, and hospitalization ward were independent predictors in readmission, the lack of follow-up, and receiving a colonoscopy. Data are represented in odds ratio (ORs) and Confidence Interval (CI) of 95%. P values < 0.05 were considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* patients affected by ALCD using a contrast-enhanced CT scan at admission undergoing NOM

Exclusion Criteria:

* immediate indication for surgery (i.e. patients with Hinchey III or IV ALCD or septic patients with Hinchey II)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients affected by ALCD
Sampling Method: Non-Probability Sample
Enrollment: 175 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Hospitalization length | one month after admission
  Comparing patients with ACLD admitted for NOM to the surgical ward with those admitted to a non-surgical ward in terms of length of stay (LOS)

SECONDARY OUTCOMES:
Follow-up and recurrences | two years after the admission
  Comparing patients with ACLD admitted for NOM to the surgical ward with those admitted to a non-surgical ward in terms of follow-up and ACLD recurrences

CONTACTS AND LOCATIONS:
Locations (1):
- Manuela Mastronardi, Trieste, TS, Italy